CLINICAL TRIAL: NCT04462263
Title: An Open-label, Single Centre, Single Oral Dose Study to Investigate the Receptor Occupancy of HTL0014242 Using [18F] FPEB in Healthy Male Subjects
Brief Title: Study to Investigate the Receptor Occupancy of HTL0014242 Using [18F] FPEB in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTL0014242-103; 2020-000602-28 (EudraCT Number); 247490 (Other: Parexel Early Phase Clinical Unit London)
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Single dose; Open-label; Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Dose HTL0014242 (Experimental): The study consists of up to 5 dosing groups, with 2 to 3 subjects per dosing group. Each subject will receive a single oral dose of HTL0014242 in the form of solid suspension capsules (1, 5, 10, and 30mg) as required. HTL0014242 will be administered in up to 5 single dose groups, with 120mg administered in the first dosing group.
  Interventions: Drug: HTL0014242

INTERVENTIONS:
Drug: HTL0014242 — Solid suspension capsule

SUMMARY:
A Study in Healthy Volunteers to Investigate How a New Drug for the Treatment of Parkinson's Disease, Dystonia and Amyotrophic Lateral Sclerosis Binds to Receptor Sites in the Brain.

DETAILED DESCRIPTION:
This is an open-label, single dose, adaptive study of orally adminstered HTL0014242 in up to 10 healthy male subjects. The primary objective is to investigate the pharmacokinetic-receptor occupancy relationship of single oral doses of HTL0014242 in healthy subjects. The secondary objectives are to assess the plasma pharmacokinetics (PK), safety and tolerability of single oral doses of HTL0014242 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, aged between 23 and 55 years inclusive, with body mass index between 18.5 and 32 kg/m2.
* Healthy on the basis of a clinical history, physical examination, electrocardiogram (ECG), vital signs and laboratory tests of blood and urine.
* Able to give fully informed consent and has suitable veins for cannulation and arterial access in both wrists
* Resting BP and heart rate within normal ranges after 5 mins rest.

Exclusion Criteria:

* Past, current or family history of mental, behavioural or neurodevelopmental disorder.
* Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, pyschiatric disorders, metabolic, allergic, dermatological, haematological, pulmonary or respiratory disorder.
* History of significant hypersensitivity, intolerance or allergy to any drug compound, food or other substance, unless approved by Investigator.
* Active neoplastic disease or history of any neoplastic disease within 5 years of screening.
* Active infection (e.g sepsis, pneumonia, abscess) or serious infection (e.g resulting in hospitalisation or requiring parenteral antibiotic treatment) within 90 days prior to dosing.
* History of stomach or intestinal surgery or resection.
* Any of following at screening or pre-dose: QT internal heart rate correction; QRS duration >120ms; PR interval > 220ms; QTc measurements/data difficult or uninterpreable; history of additional risk factors for torsades de pointe.
* drug or alcohol abuse in last 2 years.
* Alcohol consumption is > 14 units per week
* Positive Urine alcohol or drug tests
* Positive HIV, Hep B, Hep C test
* Aspartate aminotransferase, Alanine aminotransferase, Gamma glutamyl transferase, Alkaline phosphatase or total bilirubin above normal upper limits
* Participation in other clinical trials of unlicensed medicines in the previous 3 months, or 7 half-lives of the medicine (whichever is longer)
* Previously dosed with HTL0014242.
* Intention to use or using medications that interfere with drug absorption, metabolism or elimination processes incl St John's Wort, 30 days prior to dosing.
* Use of ketamine, amphetamines or MDMA with 9o days prior to dosing
* Use or intend to use any prescription or non-prescription medications within 14 days or 5 half-lives of medication, prior to dosing. Investigator and study team to determine implications on safety or study procedures, on a case-by-case basis.
* Received live attenuated vaccination within 6 weeks prior to Screening, or intends to receive vaccination during the study.
* Smoker or user of tobacco- or nicotine-containing products.
* Receipt of blood products within 2 months prior to dosing. Donation of blood / comparable blood loss 3 months prior to dosing.
* Abnormal Allen's circulation test result. Evaluation of arterial access indicates risk of occlusion or insufficient supply. Evaluation of venous access indicates difficulties in obtaining venous blood.
* Subject unable or unwilling to abstain from alcohol or caffeine-containing foods and beverages. Significant consumption of any foods or beverages containing CYP1A2 inducers with 2 weeks prior to Admission (Investigator opinion).
* Significant consumption of any foods or beverages containing Seville-type oranges, grapefruit, or poppy seeds within 7 days prior to baseline PET and admission (Investigator opinion).
* Subject, in opinion of Investigator should not participate in this study. Reply from GP, for this specific study probing psychiatric history must be received before dosing.
* Participation in research study or other radiation exposure (e.g workplace) which in conjunction with this study will exceed ionisation radiation exposure over 10mSv within 12 months prior to the Screening visit.
* Contraindication for MRI, assessed by standard pre-MRI questionnaire, that preclude subject undergoing MRI scans.
* Subject suffers from claustrophobia (incapable of undergoing MRI or PET scan) or needle phobia.
* Subject has abnormal findings per structural MRI scan at screening.

Ages: 23 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Receptor Occupancy Endpoint | Day 1 post-dose timepoint
  The regional brain Receptor Occupancy profile of HTL0014242, measured by Positron Emission Tomography (PET) imaging with[18F]FPEB
Receptor Occupancy Endpoint | Day 2 post-dose timepoint
  The regional brain Receptor Occupancy profile of HTL0014242, measured by Positron Emission Tomography (PET) imaging with[18F]FPEB

SECONDARY OUTCOMES:
Cmax: Maximum plasma concentration | Baseline up to 14(+3) days post dose
  Pharmacokinetics
Area under the plasma-concentration curve | Baseline up to 14(+3) days post dose
  Pharmacokinetics
Time to Maximum plasma concentration (Tmax) of HTL0014242 | Baseline up to 14(+3) days post dose
  Pharmacokinetics
Half-life (t1/2) of HTL0014242 | Baseline up to 14(+3) days post dose
  Pharmacokinetics
Apparent total plasma clearance (CL/F) | Baseline up to 14(+3) days post dose
  Pharmacokinetics
Incidence of Treatment Emergent Adverse Events (TEAEs) | Baseline up to 14(+3) days post dose
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No